CLINICAL TRIAL: NCT02120092
Title: The Effect of Clopidogrel and Ticagrelor With and Without Acetylsalicylic Acid (ASA) on Hemostatic System Activation at the Site of Plug Formation in Vivo in Man
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sabine Eichinger, Ao. Univ. Prof. Sabine Eichinger, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ClopidogrelTicagrelorASA
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS, Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clopidogrel + ASA (Active Comparator)
  Interventions: Drug: Clopidogrel; Drug: ASA
- Clopidogrel + Placebo (Placebo Comparator)
  Interventions: Drug: Clopidogrel; Drug: Placebo
- Ticagrelor + ASA (Active Comparator)
  Interventions: Drug: Ticagrelor; Drug: ASA
- Ticagrelor + Placebo (Placebo Comparator)
  Interventions: Drug: Ticagrelor; Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — 1x Loading dose 600 mg 6x maintenance dose 150 mg
  Arms: Clopidogrel + ASA; Clopidogrel + Placebo
Drug: Ticagrelor — 1x Loading dose: 180 mg 6x Maintenance dose: 90 mg bid
  Arms: Ticagrelor + ASA; Ticagrelor + Placebo
Drug: ASA — 7x 100mg acetylsalicylic acid (clopidogrel arm)
  1x 300 mg acetylsalicylic acid (ticagrelor arm)
  Arms: Clopidogrel + ASA; Ticagrelor + ASA
Drug: Placebo — 7x 300mg acetylsalicylic acid placebo
  Arms: Clopidogrel + Placebo; Ticagrelor + Placebo

SUMMARY:
Background: Coronary heart disease is the most common cause of death in industrialized countries. Revascularisation by percutaneous coronary angioplasty or thrombolysis is the main principle for treatment of the acute coronary syndrome. To inhibit platelet activity patients are routinely given acetylsalicylic acid (ASA) and clopidogrel, a second-generation thienopyridine. Recently, ticagrelor, a novel cyclopentyl-triazolo-pyrimidine with several pharmacological advantages, has demonstrated greater efficacy but a higher bleeding risk than clopidogrel. Coronary thrombus formation is a complex process and the antithrombotic mechanisms of platelet function inhibitors are incompletely understood. Studies in venous blood or in vitro do not truly reflect the in vivo circumstances as they often do not take into account flow conditions or the interaction between endothelium, blood cells and coagulation factors. Results from animal models may not be relevant for the prothrombotic mechanisms in humans. We have developed a technique that allows investigating hemostatic system activation directly at the site of thrombus formation in vivo in humans.

Aim: to compare the inhibitory effects of clopidogrel and ticagrelor (with and without concomitant ASA) on hemostatic system activation under circumstances close to the in vivo situation.

Design, patients and interventions: prospective, randomized, double-blind, placebo controlled parallel-group study with a 2x2 factorial design including 112 healthy volunteers who will be randomised to 4 treatment arms: ticagrelor or clopidogrel + placebo, ticagrelor or clopidogrel + ASA.

Outcome variables: Indicators of platelet and coagulation activation [ß-thromboglobulin and thromboxane B2 as well as prothrombin fragment F1+2 and D-Dimer, respectively] will be measured before and at several time points during a 8 day period in venous blood and in blood emerging from a standardized injury of the microvasculature to determine bleeding time (shed blood).

Statistical considerations: Sample size calculation is based on the percent change in the main outcome variable "β-TG in shed blood" from baseline to 2 hours after treatment start. Statistical analysis is based on the full analysis set, including all randomized subjects who received at least the starting dose of the study medication and for whom blood collections at baseline and at 2 hours after treatment start have been performed.

ELIGIBILITY:
Inclusion Criteria:

* young, healthy males

Exclusion Criteria:

* history of bleeding
* any medication
* known intolerance to study drug(s)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ß-Thromboglobulin in shed blood 2h after first study drug intake | 2 hours after first study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Eichinger-Hasenauer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria